CLINICAL TRIAL: NCT02177201
Title: Effect of Intravenous Crystalloid Volume on Postoperative Nausea and Vomiting After Tonsillectomy and/or Adenoidectomy: a Prospective, Randomized, Controlled Study
Brief Title: Effect of Intraoperative Crystalloid Volume on Postoperative Vomiting
Acronym: EICVPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Associate Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2013/255
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Sham Comparator): intravenous administration of 10 ml/kg/h 0.9% saline solution
  Interventions: Other: Group 1
- Group 2 (Active Comparator): intravenous administration of 20 ml/kg/h 0.9% saline solution
  Interventions: Other: Group 2

INTERVENTIONS:
Other: Group 1 — Intravenous access was established and 10 ml/kg/h 0.9% saline solution was delivered following the induction of anesthesia and until the end of the operation.
  Arms: Group 1
Other: Group 2 — Intravenous access was established and 20 ml/kg/h 0.9% saline solution was delivered following the induction of anesthesia and until the end of the operation.
  Arms: Group 2

SUMMARY:
Postoperative nausea and vomiting is very common in children undergone tonsillectomy and/or adenoidectomy. The purpose of this clinical trial is to evaluate the antiemetic effect of super-hydration with 0.9% saline in children undergoing specifically elective otorhinolaryngological surgery. Fluid intake reduces vomiting as seen following extended period of fasting that interrupts the perfusion in gut. Based on this knowledge, we hypothesized that administration of supplemental fluid would reduce the incidence of postoperative vomiting.

DETAILED DESCRIPTION:
At the initiation of the study, 160 patients we enrolled consecutively . Six of the patients were excluded according to the inclusion/exclusion criteria. Remaining one hundred fifty four were American Society of Anesthesia (ASA) I-II classified children , aged 2-15 yr, undergoing elective tonsillectomy, with or without adenoidectomy, under general anesthesia . Induction and maintenance of anesthesia were standardized with fentanyl, lidocaine, rocuronium and sevoflurane in nitrous oxide (N(2)O). Subjects were assigned to two groups administered with saline solution (%0.9 saline) at different rates; either 10 ml/kg/h or 20ml/kg/h delivery arms.

ELIGIBILITY:
Inclusion Criteria:ASA physical status I or II

* Age 2-15 yr
* Scheduled for elective tonsillectomy and/or adenotonsillectomy

Exclusion Criteria:

* History of diabetes
* History of mental retardation
* Obesity (BMI = > 95th percentile for age and sex)
* Intake of antiemetic or psychoactive medication within 24 hours before surgery
* Known gastroesophageal reflux

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SİNAN YILMAZ, MD, Study Director — Adnan Menderes University,Faculty of Medicine, Department of Anesthesia
Locations (2):
- Turkey (Türkiye) (2):
  - Adnan Menderes University Training and Research Hospital, Aydin, Aydın
  - Adnan Menders University, Aydin

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Intravenous 10 ml/kg/h 0.9% saline solution
- Group 2: Intravenous 20 ml/kg/h 0.9% saline solution
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 80 | 80
Completed | 77 | 77
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80 | 80 | 160
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 40 | 40 | 80
Region of Enrollment [Number; unit: participants]
  Turkey | 80 | 80 | 160
Supplemental fluid administration for vomiting [Number; unit: participants] | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Vomiting
Description: Presence of at least one episode of vomiting within the first 24 hours of postoperative is positive for definition
Time Frame: First 24 hours postoperative
Measure: Number; unit: participants
Groups:
- 10 ml/kg/h 0.9 %Saline Solution: Group 1, intravenous 10 ml/kg/h 0.9% saline solution ,
  0.9 % saline solution: After induction, IV access was established and children were randomly allocated to receive Group 1, 10 ml/kg/h 0.9% saline solution ;
- 20 ml/kg/h 0.9% Saline Solution: Group 2, intravenous 20 ml/kg/h 0.9% saline solution
  0.9 saline solution : After induction , IV access was established and children were randomly allocated to receive: 20 ml/kg/h 0.9% saline solution during intraoperatively
Arm/Group | 10 ml/kg/h 0.9 %Saline Solution | 20 ml/kg/h 0.9% Saline Solution
Number analyzed (Participants) | 77 | 77
participants
  vomiting | 11 | 9
  not vomiting | 66 | 68
Statistical Analysis 1: Comparison: 10 ml/kg/h 0.9 %Saline Solution vs 20 ml/kg/h 0.9% Saline Solution; Null hypothesis: The antiemetic effect was not significantly different for two groups in this study; Test type: Superiority or Other; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: 10 ml/kg/h 0.9 %Saline Solution vs 20 ml/kg/h 0.9% Saline Solution; 77 patients was needed in each groups for an 20% effect size, 5% alpha and 80% statistical power for postoperative vomiting; Test type: Superiority or Other; p < 0.05, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: No adverse event were detected for all participants in the first 24 hours.
Description: No adverse event were detected for all participants in the first 24 hours.
Groups:
- Group 1 Intravenous 10ml/kg/h 0.9 %Saline Solution: Group 1, intravenous 10 ml/kg/h 0.9% saline solution , After induction, IV access was established and children were randomly allocated to receive one of two interventions: Group 1, 10 ml/kg/h 0.9% saline solution ; Group 2, 20 ml/kg/h 0.9% saline solution by intravenous during intraoperatively. In both groups no adverse events were observed.
- Group 2 Intravenous 20ml/kg/h 0.9 %Saline Solution: Group 2, intravenous 20 ml/kg/h 0.9% saline solution. After induction, IV access was established and children were randomly allocated to receive one of two interventions: Group 1, 10 ml/kg/h 0.9% saline solution ; Group 2, 20 ml/kg/h 0.9% saline solution by intravenous during intraoperatively. In both groups no adverse events were observed.
Arm/Group | Group 1 Intravenous 10ml/kg/h 0.9 %Saline Solution | Group 2 Intravenous 20ml/kg/h 0.9 %Saline Solution
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes